CLINICAL TRIAL: NCT06689527
Title: An Open-label, Single-arm Study to Evaluate the CYP3A4 Induction Potential of Vamorolone on the Pharmacokinetics of Midazolam (a Sensitive CYP3A4 Probe) in Healthy Subjects.
Brief Title: Evaluation of Vamorolone CYP3A4 Induction on Midazolam (a Sensitive CYP 3A4 Substrate) Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Santhera Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SNT-I-VAM-025; 2024-513845-36-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-05; First posted 2024-11-14 (Actual); Results first posted 2025-12-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Drug Interaction
Keywords: Drug-Drug-Interaction Study
MeSH Terms: interventions — VBP15 compound; Drug Evaluation; Midazolam

STUDY DESIGN:
Intervention Model Description: A single-center, open-label, single-arm, fixed-sequence, design. Healthy male and female subjects (18 to 55 years, inclusive) are eligible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Midazolam/Vamorolone (Experimental): Single oral dose midazolam 2.5mg on day 1 Single oral suspension vamorolone 6mg/kg on day 3 to day 13 Single oral dose midazolam 2.5mg + Single oral suspension vamorolone 6mg/kg on day 14
  Interventions: Drug: Vamorolone; Drug: Midazolam

INTERVENTIONS:
Drug: Vamorolone — Days 3 to 14: 6 mg/kg vamorolone once daily.
  Other Names: Test Drug
Drug: Midazolam — Day 1 and 14: Single oral doses of 2.5 mg midazolam
  Other Names: Reference Drug

SUMMARY:
The purpose of this study was to investigate how vamorolone affects the CYP3A4 enzyme in humans by measuring the pharmacokinetics of midazolam and its metabolite, 1'-hydroxymidazolam, in healthy subjects. The pharmacokinetics of midazolam were measured on Day 1 and then on Day 14 to investigate the potential interaction between the two compounds.

The safety and the tolerability was also investigated.

DETAILED DESCRIPTION:
This was a non-randomized, single-center, open-label, single-sequence, single-arm Phase I study.

* Day 1: Participants received a single dose of 2.5 mg midazolam in fasted state in the morning.
* Day 2: Wash-out period.
* Days 3 to 13: Participants received daily doses of 6 mg/kg vamorolone in the morning within 30 minutes after start of a standard breakfast.
* Day 14: Participants received single doses of 2.5 mg midazolam and 6 mg/kg vamorolone in fasted state in the morning.
* Safety and tolerability parameters were collected during the entire study phase from screening to follow-up.
* Blood samples for PK assessment of midazolam and 1'-hydroxymidazolam were collected from predose through 10 hours following the midazolam doses on Days 1 and 14.
* Blood samples for PK assessment of vamorolone were collected throughout the vamorolone dosing period.
* Blood and urine biomarkers samples for CYP3A4 induction assessment were collected throughout the treatment period.
* On Day 28, a follow-up safety phone call was done

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 to 55 years inclusive, at the time of signing the informed consent.
2. Subject is overtly healthy as determined by medical evaluation including medical history, physical examination, vital signs, laboratory tests, and ECG.
3. Body weight ≥ 50 kg and a BMI ≥ 18 kg/m2 and ≤ 29.9 kg/m2 at screening.
4. Male and female. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male subjects:

   • If the subject is a sexually active man and not surgically sterilized, he must be willing to:
   * Abstain from sexual intercourse or
   * Use a condom plus another form of contraception, (e.g., spermicide, IUD, birth control pills taken by female partner) if engaging in sexual intercourse with a woman who could become pregnant.
   * Use a condom during sexual intercourse with pregnant or lactating women.
   * Must not father a child and must refrain from donating sperm from administration of the first dose and up to 3 months after the last dose of study treatment.

   Female subjects:

   All women (regardless of their status, i.e. WOCBP and WONCBP; for definitions see Section 10.4.1) must have a negative serum β-hCG pregnancy test prior to the initiation of the study treatments. FSH levels of suspected postmenopausal females must be > 30 mIU/mL.

   Vamorolone has the potential to induce CYP3A4, which may result in a reduction in the effectiveness of contraceptives that are metabolized by CYP3A4 such as hormonal contraceptives when co-administered with vamorolone. Therefore, hormonal contraceptives by any route of administration are contraindicated.

   Women participating in the study must be either:
   * WONCBP or
   * WOCBP using, during the length of the study and for at least 3 months after the stop of the study treatments, 1 of the following contraceptive methods plus a condom:

     * IUD during the study and up to 3 months after the last administration of the study treatments
     * Any IUD with published data showing that the lowest expected failure rate is less than 1% per year (not all IUDs meet this criteria)
     * Any other methods with published data showing that the lowest expected failure rate for birth control is less than 1% per year, or
     * Abstinent from intercourse for 2 weeks before exposure to the study treatments, throughout the clinical trial until 3 months following discontinuation of the study treatments, or
     * Have a male partner who is sterile prior to the woman's entry into the study and is the sole sexual partner for that woman during the study period.

   The Investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with an early undetected pregnancy.
5. Subject is a non-smoker for at least 3 months prior exposure to the study treatments. Subject must also have abstained from use of other nicotine containing products (e.g., nicotine patch, chewing gum or e-cigarettes) for at least 3 months before exposure to the study treatments.
6. Capable of giving signed informed consent as described in Section 10.1, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol prior to any clinical study specific procedure.
7. Supine systolic blood pressure ≥ 90 mmHg and ≤ 140 mmHg; diastolic blood pressure ≥ 50 mmHg and ≤ 90 mmHg and pulse rate ≥ 45 bpm and ≤ 90 bpm, and tympanic body temperature ≥ 35.0 °C and ≤ 37.5 °C at screening.
8. Subjects must be able to communicate well with the Investigator and comply with the protocol requirements, instructions, and protocol related restrictions (e.g. dietary, fluid and lifestyle restrictions from screening to study completion; Section 5.3).
9. Subjects must be able to swallow the study treatments as per protocol.

   Exclusion Criteria:
10. A past medical history of clinically significant abnormalities or a history/family history of long QT interval syndrome, structural cardiac abnormalities (including but not limited to hypertrophic cardiomyopathy, valvulopathy, and congenital defects), or cardiogenic syncope.
11. An abnormal ECG, defined as:

    * PR > 215 msec and < 100 msec, QRS complex > 120 msec; QTcF > 450 msec by automated reading
    * Any clinically significant ST/T wave abnormalities
    * Any atrial or ventricular arrhythmias
12. A past medical history of myocardial infarction, angina pectoris, atherosclerosis or other clinically significant heart disease (e.g., congestive heart failure, uncontrolled hypertension, history of labile hypertension).
13. A past medical history of peptic ulcers, diverticulitis, and non-specific ulcerative colitis.
14. History of complaints of frequent dizziness and /or vomiting spells or lightheadedness ("frequent" defined as incidence occurs more than once every week) or history of/or present sleep apnea.
15. Any history or evidence of any clinically relevant, gastrointestinal, respiratory, hepatic, renal, endocrinologic, hematologic, immunologic, metabolic, genitourinary, pulmonary, neurologic, dermatologic, musculoskeletal, and/or other major disease or malignancy as determined by medical evaluation (including physical examination) capable of significantly altering the absorption, metabolism, or elimination of drugs; constituting a risk when taking the study treatments; or interfering with the interpretation of data.
16. Known Gilbert's syndrome.
17. Any clinically relevant history of allergic conditions requiring hospitalization or prolonged systemic treatment (including drug allergies, allergic asthma, eczema, allergies requiring therapy with corticosteroids or anaphylactic reactions); but excluding untreated, asymptomatic, seasonal allergies at time of dosing or allergic contact sensitizations (e.g., nickel allergy).
18. Known or suspected hypersensitivity or contraindications to vamorolone and/or midazolam or any components of the formulation used.
19. Relevant current acute or chronic/recurrent viral, bacterial, fungal, or parasitic infections (e.g., pulmonary/upper respiratory, gastrointestinal, urinary, skin, or ENT infections) at screening or within 28 days prior to administration of the study treatments.
20. Use of any concomitant medication or any drugs / medicines (including dietary supplements, natural and herbal remedies, and hormone replacement therapy) within 2 weeks or 5 times the half-life of the respective drug, whichever is longer, prior to the first administration of the study treatments.

    Occasional use of paracetamol up to 2 g/day or ibuprofen up to 1.2 g/day (medicinal products in their original packaging, approved and marketed in Germany) is permitted.

    Oral, injectable, and implantable contraceptives as outlined in Section 5.1 are permitted.
21. Previous exposure to vamorolone.
22. Any use of corticoids within 6 months prior to the first administration of the study treatments.
23. Administration of live, attenuated, replication-competent vaccines within 6 weeks prior to the first administration of the study treatments until 2 weeks after the follow-up visit. Administration of vector-based or mRNA COVID-19 vaccines within 2 weeks prior to the first administration of the study treatments until 2 weeks after the follow-up visit.
24. Treatment with biologic agents (such as monoclonal antibodies including marketed drugs) within 3 months or 5 half-lives (whichever is longer) prior to the first administration of the study treatments.
25. Use of any investigational drug or participation in any clinical study within 30 days or 5 half-lives (whichever is longer) prior to the expected date of first administration of study treatments or planning to take other investigational drugs during the study.
26. Positive results for HBsAg, anti-HCV, anti-HIV 1 and 2, and HIV 1-p24 antigen at screening.
27. Positive screen for alcohol, drugs of abuse and cotinine at screening.
28. Elevations in ALT > 1.1 x ULN, AST > 1.2 x ULN, serum bilirubin > 1.2 x ULN, creatinine > 1.1 x ULN and and HbA1c > ULN at screening. A case-by-case decision for any abnormality must be discussed with the Sponsor before inclusion.
29. TSH outside of normal ranges.
30. eGFR based on the CKD-EPI (details for calculation see Section 10.2) of < 90 mL/min at screening.
31. Potassium or magnesium blood concentration below the lower limit of normal at screening.
32. Subjects who are unwilling to adhere to contraceptive requirements.
33. Higher than low-risk alcohol consumption i.e., consumption of an average weekly alcohol intake of > 21 units/week for men and > 14 units/week for women. 1 unit (12 g) corresponds to 0.3 L of beer/day or 0.12 L of wine/day or 1 glass (at 2 cL) of spirits/day.
34. Excessive consumption of caffeine- or xanthine-containing food or beverages (> 5 cups of coffee a day or equivalent) or inability to stop consuming from 48 hours prior to first planned administration of study treatments.
35. Consumption of alcohol from 48 hours prior to admission.
36. Consumption of high dose resveratrol-containing products or products with enzyme-inducing or enzyme-inhibiting properties (for details refer to Section 5.3.1) 14 days prior to first administration of study treatment.
37. Regular consumption of poppy seed containing food prior to first administration of study treatment.
38. Any use of drugs-of-abuse or alcohol abuse within 1 month prior to dosing.
39. Subject with vegetarian, vegan, or restricted diet (e.g., gluten-free) or not willing or able to eat the complete standard meals.
40. Female subject who has been pregnant within 6 months prior to screening or breastfeeding or lactating within 3 months prior to screening or plans to become pregnant during the clinical study period and for 3 months after final study treatment administration.
41. Donation or loss of more than 400 mL of blood or received a transfusion of any blood or blood products within 30 days, or donated plasma within 30 days prior to first administration of study treatment.
42. Strenuous physical activity within 72 h to admission.
43. Employee of the Sponsor, the Nuvisan Group, or other Contract Research Organization involved in the clinical study.
44. Legal incapacity or limited legal capacity, or incarceration and vulnerable subjects.
45. Inability to understand or communicate reliably with the Investigator or considered by the Investigator to be unable to or unlikely to co-operate with the protocol requirements, instructions, and study-related restrictions.
46. History of non-compliance to medical regimens and subjects who are considered potentially unreliable (e.g., refuse to comply with study regulations).
47. Any other conditions or factors which in the opinion of the Investigator may interfere with study conduct.
48. Changes in medical conditions compared to screening, as judged by the Investigator.
49. Body weight < 50 kg.
50. Changes in prior/concomitant therapy compared to screening, as judged by the Investigator.
51. Positive screen for alcohol, drugs of abuse and cotinine test upon admission.
52. Changes in other exclusion criteria compared to screening, as judged by the Investigator.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2024-08-13 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lissy, MD, Principal Investigator — Nuvisan GmbH
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

RESULTS

PARTICIPANT FLOW:
Groups:
- Vamorolone/Midazolam: both Test Drug and Reference Drug are administered in this arm
  Vamorolone: Days 3 to 14: 6 mg/kg vamorolone once daily.
  Midazolam: Day 1 and 14: Single doses of 2.5 mg midazolam
Period: Overall Study
Arm/Group | Vamorolone/Midazolam
Started | 18
Completed | 18
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Vamorolone/Midazolam: both Test Drug (vamorolone) and Reference Drug (midazolam) are administered in this arm
  Vamorolone: Days 3 to 14: 6 mg/kg vamorolone once daily.
  Midazolam: Day 1 and 14: Single oral doses of 2.5 mg midazolam
Arm/Group | Vamorolone/Midazolam
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (9.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Germany | 18
Height [Mean (Standard Deviation); unit: cm] | 170.5 (10.55)
Weight [Mean (Standard Deviation); unit: kg] | 69.34 (10.876)
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index
  kg/m2 | 23.81 (2.389)
Premenopausal/Postmenopausal Status [Count of Participants; unit: Participants] — This measure only concerned female participants in the study and provides the number of those who were premenopausal or postmenopausal. Population: This population only includes female participants.
  Participants
    number analyzed (Participants) | 10
    Premenopausal Status | 8
    Postmenopausal Status | 2

OUTCOME MEASURES:

1. Primary Outcome: AUC0-tlast of Midazolam
Description: Area under the plasma concentration-time curve from 0 to the time of the last observed concentration (h*pg/mL) on day 1 and day 14. The timepoints at which the data were collected to create the curve are as follows: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours postdose.
Time Frame: Day 1 and Day 14
Population: PK Set - Midazolam: a subset of the Safety Set and includes all subjects who completed the scheduled vamorolone and midazolam dosing and provided an evaluable midazolam PK profile on at least one of the following days Day 1 and Day 14. No vomiting should occur within 4 hours following midazolam and/or vamorolone administration.
  This PK set was used for PK concentration summary and PK parameter summary for midazolam and 1'-hydroxymidazolam.
Measure: Mean (Standard Deviation); unit: h*pg/ml
Groups:
- Midazolam Alone on Day 1: Day 1: Single oral of midazolam dose 2.5 mg
- Midazolam Co-administered With Vamorolone on Day 14.: Day 14: Single oral midazolam dose of 2.5mg + Single oral suspension vamorolone dose of 6mg/kg
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h*pg/ml | 34331.8 (11854.73) | 28619.6 (11447.17)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subjects as random effect; Test type: Other; Ratio of Geometric LS Mean (%) = 83.95, 90% CI 2-sided [74.08 to 93.59] — The linear mixed model was applied to log-transformed PK parameter AUC0-tlast, of midazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

2. Primary Outcome: AUC0-inf of Midazolam
Description: Area under the plasma concentration-time curve from zero to infinite time on day 1 and day 14. The timepoints at which the data were collected to create the curve are as follows: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours postdose and extrapolation to infinity.
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*pg/mL
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 17
h*pg/mL | 38028.2 (14556.59) | 30337.7 (12238.52)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subjects as random effect; Test type: Other; Ratio of Geometric LS Mean ( = 83.05, 90% CI 2-sided [74.18 to 95.00] — The linear mixed model was applied to log-transformed PK parameter AUC0-inf of midazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

3. Primary Outcome: Cmax of Midazolam
Description: maximum measured concentration of midazolam after administration of midazolam until the last collection time, i.e., 10 hours after dosing on day 1 and day 14
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
pg/ml | 15704 (5495.3) | 13875 (4995.2)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subject as random effect; Test type: Other; Ratio of Geometric LS Mean (%) = 88.59, 90% CI 2-sided [79.44 to 98.79] — The linear mixed model was applied to log-transformed PK parameter Cmax of midazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

4. Primary Outcome: AUC0-tlast of 1'-Hydroxymidazolam
Description: as for outcome 1
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*pg/ml
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h*pg/ml | 11019.7 (4377.21) | 12669.0 (5085.13)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subject as random effect; Test type: Other; Ratio of Geometric LS Mean (%) = 114.55, 90% CI 2-sided [101.59 to 129.18] — The linear mixed model was applied to log-transformed PK parameter AUC0-tlast of 1'-hydroxymidazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

5. Primary Outcome: AUC-inf of 1'-Hydroxymidazolam
Description: Area under the plasma concentration-time curve from 0 to the infinite time (h*pg/mL) on day 1 and Day 14. The timepoints at which the data were collected to create the curve are as follows: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 10 hours postdose and extrapolation to infinity.
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*pg/ml
Groups:
- Midazolam Alone on Day 1: Day 1: Single oral of miazolam dose 2.5 mg
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h*pg/ml | 11592.1 (4592.86) | 13211.4 (5225.69)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subject as random effect; Test type: Other; Ratio of Geometric LS Mean (%) = 113.70, 90% CI 2-sided [101.29 to 127.63] — The linear mixed model was applied to log-transformed PK parameter AUC0-inf, of 1'-hydroxymidazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

6. Primary Outcome: Cmax of 1'-Hydroxymidazolam
Description: maximum measured concentration of 1'-Hydroxymidazolam after administration of midazolam until the last collection time, i.e., 10 hours after dosing
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
pg/ml | 5846 (2748.8) | 7920 (3988.6)
Statistical Analysis 1: Comparison: Midazolam Alone on Day 1 vs Midazolam Co-administered With Vamorolone on Day 14; Linear model with treatment as fixed effect and subject as random effect; Test type: Other; Ratio of Geometric LS Mean (%) = 128.67, 90% CI 2-sided [105.36 to 157.13] — The linear mixed model was applied to log-transformed PK parameter Cmax of 1'-hydroxymidazolam based on the PK Set to assess treatment differences on the log scale of midazolam with vamorolone vs midazolam alone (Day 14 vs Day 1)

7. Secondary Outcome: Tmax of Midazolam
Description: Time to reach observed maximal concentration of midazolam after administration of midazolam until the last collection time, i.e., 10 hours after administration on day 1 and day 14
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h | 0.500 [0.25 to 1.52] | 0.500 [0.25 to 2.02]

8. Secondary Outcome: CL/F of Midazolam
Description: The apparent clearance measures how quickly a drug leaves the body, considering how much reaches it after being taken orally. It was calculated using the formula: Dose/AUCinf on day 1 and day 14. The timepoints used were as follows: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours on day 1 and day 14
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 17
L/h | 78.80 (45.683) | 93.27 (31.471)

9. Secondary Outcome: Vz/F of Midazolam
Description: Vz/F is the ratio of the volume of distribution of a drug to its bioavailability. It describes how widely the drug is distributed in the body after oral administration. It was calculated based on the terminal phase (ℷz)using the formula: Dose /ℷz.AUCinf on day 1 and day 14. The timepoints were as follows: predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours.
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 17
L | 311.0 (110.54) | 414.3 (123.97)

10. Secondary Outcome: t1/2 of Midazolam
Description: Elimination half-life is the amount of time it takes for the concentration of the drug (midazolam) in the body to decrease by half after administration on day 1 and day 14. The collection times were predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours.
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h | 2.980 (0.7003) | 3.305 (0.8752)

11. Secondary Outcome: Tmax of 1'-Hydroxymidazolam
Description: Time to reach observed maximal concentration of 1'-Hydroxymidazolam after administration of midazolam until the last collection time, i.e., 10 hours after dosing on day 1 and day 14
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h | 0.500 [0.25 to 1.52] | 0.500 [0.50 to 2.02]

12. Secondary Outcome: t1/2 of 1'-Hydroxymidazolam
Description: Elimination half-life is the amount of time it takes for the concentration of the drug (1'-Hydroxymidazolam) in the body to decrease by half on day 1 and day 14. The collection times were predose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10 hours.
Time Frame: Day 1 and Day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Midazolam Alone on Day 1 | Midazolam Co-administered With Vamorolone on Day 14.
Number analyzed (Participants) | 18 | 18
h | 2.215 (0.4131) | 2.122 (0.3770)

13. Secondary Outcome: Predose Concentration (Ctrough) of Vamorolone
Description: Concentration measurements taken just before the first administration of vamorolone on day 3, and at the end of each vamorolone dosing interval before the next dose on days 4, 7, 11, 13, and 14.
Time Frame: Day 3, Day 4, Day 7, Day 11, Day 13, Day 14
Population: PK-Set Vamorolone: This analysis set is a subset of the safety set and includes all subjects who completed at least one scheduled vamorolone dose without vomiting within 4 hours immediately following that vamorolone administration and provided at least one valid PK concentration data for vamorolone.
  This PK set was used for PK concentration summary and PK parameter summary for vamorolone
Measure: Mean (Standard Deviation); unit: ng/ml
Groups:
- Vamorolone Alone on Day 4; Vamorolone Alone on Day 7; Vamorolone on Day 11; Vamorolone Alone on Day 13: Oral suspension of vamorolone 6 mg/kg
- Vamorolone Coadministrated With Midazolam on Day 14: Oral suspension of vamorolone 6 mg/kg coadministrated with single oral of midazolam dose 2.5 mg
Arm/Group | Vamorolone Alone on Day 4 | Vamorolone Alone on Day 7 | Vamorolone on Day 11 | Vamorolone Alone on Day 13 | Vamorolone Coadministrated With Midazolam on Day 14
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18
ng/ml | 9.397 (20.182) | 3.486 (5.0864) | 3.816 (5.1055) | 2.070 (2.5436) | 1.303 (1.5972)

14. Secondary Outcome: Urinary 6β-hydroxycortisol to Cortisol Ratio
Description: Urinary 6β-hydroxycortisol to cortisol ratio is used as in vivo biomarkers for CYP3A4 activity. The impact of vamorlone on adrenal suppression could result in alterations in urinary cortisol and 6-β-hydroxycortisol levels.. Thus, the 6-β-hydroxycortisol to cortisol ratio is an unreliable measure of vamorolone's CYP3A4 induction potential.
Time Frame: Day 1, Day 3, Day 4, Day 7, Day 11, Day 14, Day 15
Population: Safety Set: All subjects assigned to study treatment and who received at least 1 dose of study treatment. Subjects were analyzed according to the treatment they actually received.
Measure: Mean (Standard Deviation); unit: ratio
Groups:
- Midazolam Alone on Day 1: Single oral midazolam dose 2.5mg
- Vamorolone Alone on Day 3; Vamorolone Alone on Day 4; Vamorolone Alone on Day 7; Vamorolone on Day 11: Oral suspension of vamorolone 6 mg/kg
- No Treatment on Day 15: No drug administration; end of study treatment
Arm/Group | Midazolam Alone on Day 1 | Vamorolone Alone on Day 3 | Vamorolone Alone on Day 4 | Vamorolone Alone on Day 7 | Vamorolone on Day 11 | Vamorolone Coadministrated With Midazolam on Day 14 | No Treatment on Day 15
Number analyzed (Participants) | 17 | 18 | 11 | 11 | 10 | 5 | 14
ratio | 3.496 (1.4406) | 2.856 (1.1187) | 4.739 (0.95864) | 5.518 (1.4118) | 5.234 (1.4441) | 5.388 (0.99344) | 6.571 (2.6256)

15. Secondary Outcome: Plasma 4β-hydroxycholesterol Level
Description: The plasma concentration of 4-β-hydroxycholesterol is used as an in vivo marker to assess CYP3A4 induction activity
Time Frame: Day 1, Day 3, Day 4, Day 7, Day 11, Day 14, Day 15
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Midazolam Alone on Day 1 | Vamorolone Alone on Day 3 | Vamorolone Alone on Day 4 | Vamorolone Alone on Day 7 | Vamorolone on Day 11 | Vamorolone Coadministrated With Midazolam on Day 14 | No Treatment on Day 15
Number analyzed (Participants) | 18 | 18 | 18 | 18 | 18 | 18 | 18
ng/ml | 40.75 (44.696) | 41.51 (34.890) | 40.36 (33.582) | 45.53 (34.426) | 38.87 (20.366) | 36.73 (19.713) | 38.93 (19.328)

ADVERSE EVENTS:
Time Frame: All AEs and SAEs were collected from signing the informed consent until the safety follow-up visit on Day 28 i.e., approximately 2 weeks after the last midazolam administration/early discontinuation visit. After the conclusion of the study, investigators did not actively seek AEs and SAEs. All SAEs had to be recorded and reported to the sponsor or designee within 24 hours. Investigators had to report any SADR (SAE considered related to the IMP) to the sponsor.
Groups:
- Vamorolone Alone on Day 3 to Day 13: Oral suspension of vamorolone 6 mg/kg
Arm/Group | Midazolam Alone on Day 1 | Vamorolone Alone on Day 3 to Day 13 | Vamorolone Coadministrated With Midazolam on Day 14
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 2/18 | 8/18 | 2/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Midazolam Alone on Day 1 (N=18) | Vamorolone Alone on Day 3 to Day 13 (N=18) | Vamorolone Coadministrated With Midazolam on Day 14 (N=18)
Fatigue (General disorders) | 1 (2) | 0 (0) | 0 (0) — 2 events reported on Day 1with mild severity and one was related to midazolam treatment
Headache (Nervous system disorders) | 0 (0) | 1 (2) | 1 (1) — 3 events of mild intensity. The first two occurred on Days 5 and 9, were unrelated to the study drug, and resolved without treatment. The third event occurred on Day 14 and was related to midazolam. The subject took 400 mg of ibuprofen.
Initial Insomnia (Psychiatric disorders) | 0 (0) | 3 (3) | 0 (0) — 3 subjects reported initial insomnia of mild intensity with a duration of 4 days. These TEAEs were assessed by the investigator as related to vamorolone. The events resolved without any concomitant medication.
ALT increased (Investigations) | 0 (0) | 1 (1) | 0 (0) — The increased ALT level peaked on Day 15 and lasted for 26 days, beginning on Day 9. It resolved without treatment. This moderate event was related to vamorolone.
Amylase increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Amylase level peaked on Day 15and resolved to normal levels by Day 21. The event seerity is moderate and was not related to study treatment
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Lipase increased with severe intensity peaked on Day 15 and resolved by Day 21 without any treatment. The event was not related to study drugs
Foreign body sensation in eyes (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — The event started on Day 11 and lasted 2 days with mild intensity. The event resolved without any treatment and was not related to the study drugs
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — The heartburn event, which was mild in intensity, started on Day 12 and was related to the vamorolone treatment, but it resolved without any treatment.
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) — A mild case of nasopharyngitis started on Day 10 and lasted for 18 days. This event was not related to the study treatment and resolved without concomitant medication.
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) — 2 events of nasal discomfort, both of mild intensity related to vamorolone and resolved without treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-06-05): https://cdn.clinicaltrials.gov/large-docs/27/NCT06689527/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/27/NCT06689527/SAP_001.pdf